CLINICAL TRIAL: NCT06393517
Title: A PHASE 1, OPEN-LABEL, RANDOMIZED, 5-PERIOD, 6-SEQUENCE, CROSSOVER STUDY TO COMPARE THE SINGLE-DOSE PHARMACOKINETICS OF IMMEDIATE-RELEASE AND MODIFIED-RELEASE FORMULATIONS OF PF-06954522 ADMINISTERED ORALLY TO HEALTHY ADULT PARTICIPANTS
Brief Title: A Study to Learn How Different Forms of the Study Medicine Called PF-06954522 Are Taken up Into the Blood in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: C4001005
Record Dates: First submitted 2024-04-26; First posted 2024-05-01 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Healthy Participants

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Sequence 1 (Experimental): Participants will receive a single dose (Dose Level 1 and 2) of PF-06954522 as:
  Formulation 1 , Formulation 2, and Formulation 3 under fasted conditions in Periods 1, 2, and 3, respectively, followed by Formulations 2 and 3 under fed conditions in Periods 4 and 5, respectively.
  Interventions: Drug: PF-06954522 IR (Formulation 1); Drug: PF-06954522 MR (Formulation 2); Drug: PF-06954522 MR (Formulation 3)
- Sequence 2 (Experimental): Participants will receive a single dose (Dose Level 1 and 2) of PF-06954522 as:
  Formulation 2, Formulation 3, and Formulation 1 under fasted conditions in Periods 1, 2, and 3, respectively, followed by Formulations 2 and 3 under fed conditions in Periods 4 and 5, respectively.
  Interventions: Drug: PF-06954522 IR (Formulation 1); Drug: PF-06954522 MR (Formulation 2); Drug: PF-06954522 MR (Formulation 3)
- Sequence 3 (Experimental): Participants will receive a single dose (Dose Level 1 and 2) of PF-06954522 as:
  Formulation 3, Formulation 1, and Formulation 2, under fasted conditions in Periods 1, 2, and 3, respectively, followed by Formulations 2 and 3 under fed conditions in Periods 4 and 5, respectively.
  Interventions: Drug: PF-06954522 IR (Formulation 1); Drug: PF-06954522 MR (Formulation 2); Drug: PF-06954522 MR (Formulation 3)
- Sequence 4 (Experimental): Participants will receive a single dose (Dose Level 1 and 2) of PF-06954522 as:
  Formulation 3, Formulation 2, and Formulation 1 under fasted conditions in Periods 1, 2, and 3, respectively, followed by Formulations 3 and 2 under fed conditions in Periods 4 and 5, respectively.
  Interventions: Drug: PF-06954522 IR (Formulation 1); Drug: PF-06954522 MR (Formulation 2); Drug: PF-06954522 MR (Formulation 3)
- Sequence 5 (Experimental): Participants will receive a single dose (Dose Level 1 and 2) of PF-06954522 as:
  Formulation 1, Formulation 3, and Formulation 2 under fasted conditions in Periods 1, 2, and 3, respectively, followed by Formulations 3 and 2 under fed conditions in Periods 4 and 5, respectively.
  Interventions: Drug: PF-06954522 IR (Formulation 1); Drug: PF-06954522 MR (Formulation 2); Drug: PF-06954522 MR (Formulation 3)
- Sequence 6 (Experimental): Participants will receive a single dose (Dose Level 1 and 2) of PF-06954522 as:
  Formulation 2, Formulation 1, and Formulation 3 under fasted conditions in Periods 1, 2, and 3, respectively, followed by Formulations 3 and 2 under fed conditions in Periods 4 and 5, respectively.
  Interventions: Drug: PF-06954522 IR (Formulation 1); Drug: PF-06954522 MR (Formulation 2); Drug: PF-06954522 MR (Formulation 3)

INTERVENTIONS:
Drug: PF-06954522 IR (Formulation 1) — Participants to receive a single dose (Dose Level 1 and 2) of PF-06954522 Formulation 1 by mouth
Drug: PF-06954522 MR (Formulation 2) — Participants to receive a single dose (Dose Level 1 and 2) of PF-06954522 Formulation 2 by mouth.
Drug: PF-06954522 MR (Formulation 3) — Participants to receive a single dose (Dose Level 1 and 2) of PF-06954522 Formulation 3 by mouth

SUMMARY:
The purpose of this study is to compare three finished products of PF-06954522 in terms of the uptake into the blood stream.

This study is seeking participants who are:

- Healthy male or female participants aged 18 years or older.

All participants in this study will receive PF-06954522 once by mouth. The participants may receive different tablets by mouth for PF-06954522.

The study will compare experiences of people receiving three different products of PF-06954522. This will help understand how much PF-06954522 is taken up into the blood for each product given.

Participants will take part into the study for about 77 days. During this time participants will have to stay onsite for 21 days. There will be one follow up (by telephone) study visit.

ELIGIBILITY:
Inclusion Criteria:

* Male and female participants of non-childbearing potential aged 18 years or older who are overtly healthy as determined by medical evaluation including medical history, physical examination, laboratory tests, vital signs, and electrocardiograms.
* Body mass index of 16-32 kg/m2; and a total body weight >50 kg (110 lbs).

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurological, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at the time of dosing).
* Personal or family history of medullary thyroid carcinoma (MTC) or multiple endocrine neoplasia type 2, or participants with suspected MTC per the investigator's judgement.
* Any medical or psychiatric condition including recent (within the past year) or active suicidal ideation/behavior or laboratory abnormality that may increase the risk of study participation or, in the investigator's judgment, make the participant inappropriate for the study.
* Use of any prohibited prior/concomitant medication(s).
* A positive urine drug test at screening or admission.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2024-04-30 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2024-09-01 (Actual)

PRIMARY OUTCOMES:
Area Under the Curve from time zero to extrapolated infinite time (AUCinf) of PF-06954522 to evaluate the relative bioavailability of three PF-06954522 formulations administered in the fasted state. | 0 hours (pre-dose) to 72 hours (extrapolated to infinite time) post PF-06954522 dose in each period
Maximum Observed Plasma Concentration (Cmax) of PF-06954522 to evaluate the relative bioavailability of three PF-06954522 formulations administered in the fasted state. | 0 hours (pre-dose) to 72 hours post PF-06954522 dose in each period

SECONDARY OUTCOMES:
Number of Participants with Treatment-Emergent Adverse Events (AEs) | From baseline up to 49 days after PF-06954522 dose in Period 1 Day 1
Number of Participants with Laboratory Test Abnormalities | From baseline up to 72 hours after PF-06954522 dose in each period
Number of Participants with Summary of Post-Baseline Vital Signs Data | From baseline up to 72 hours after PF-06954522 dose in each period
Number of Participants who met Defined Electrocardiogram (ECG) Criteria | From baseline up to 72 hours after PF-06954522 dose in each period
Area Under the Curve from time zero to extrapolated infinite time (AUCinf) of PF-06954522 to evaluate the relative bioavailability of two PF-06954522 formulations administered in the fed state compared to fasted state. | 0 hours (pre-dose) to 72 hours (extrapolated to infinite time) post PF-06954522 dose in each period
Maximum Observed Plasma Concentration (Cmax) of PF-06954522 to evaluate the relative bioavailability of two PF-06954522 formulations administered in the fed state compared to the fasted state. | 0 hours (pre-dose) to 72 hours post PF-06954522 dose in each period

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (2):
- United States (2):
  - Pfizer Clinical Research Unit - New Haven, New Haven, Connecticut
  - Pfizer Clinical Research Unit, New Haven, Connecticut

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C4001005